CLINICAL TRIAL: NCT02899221
Title: Phase I Study of Hyperthermia Combined With High Dose Rate Salvage Radiotherapy for the Treatment of Radiation Recurrent Prostate Cancer
Brief Title: Hyperthermia and High Dose Rate Radiation Therapy in Treating Patients With Recurrent Prostate Cancer After Radiation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16D.246; JT 8400 (Other: JeffTrial Number)
Record Dates: First submitted 2016-09-08; First posted 2016-09-14 (Estimated); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Recurrent Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Brachytherapy; Diathermy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (high dose rate brachytherapy, hyperthermia) (Experimental): Patients undergo high dose rate brachytherapy for 15-30 minutes. Immediately after radiation therapy (no longer than 90 minutes), patients undergo interstitial hyperthermia treatment for up to 60 minutes.
  Interventions: Radiation: High-Dose Rate Brachytherapy; Procedure: Hyperthermia Treatment; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Radiation: High-Dose Rate Brachytherapy — Undergo high dose rate brachytherapy
  Other Names: Brachytherapy; High Dose; HDR; High dose brachytherapy (procedure)
Procedure: Hyperthermia Treatment — Undergo interstitial hyperthermia treatment
  Other Names: Clinical Hyperthermia; Diathermy; Hyperthermia; Hyperthermia Therapy
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best way to give hyperthermia and high dose rate radiation therapy in treating patients with prostate cancer that has come back after prior radiation treatment. Radiation therapy, such as high dose rate brachytherapy, uses radioactive material placed directly into or near a tumor to kill tumor cells. Hyperthermia therapy may make tumor cells more sensitive to the effects of radiation therapy by heating them to several degrees above normal body temperature. Giving hyperthermia and high dose rate radiation therapy may work better in treating patients with recurrent prostate cancer after radiation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and feasibility of combined single fraction high dose rate (HDR) brachytherapy followed immediately by interstitial hyperthermia treatment of radio-recurrent prostate cancer.

SECONDARY OBJECTIVES:

I. To assess long-term toxicity. II. To provide a preliminary assessment of efficacy. III. To obtain blood for future analysis of immune response to combined radiation therapy and hyperthermia.

OUTLINE:

Patients undergo high dose rate brachytherapy for 15-30 minutes. Immediately after radiation therapy (no longer than 90 minutes), patients undergo interstitial hyperthermia treatment for up to 60 minutes.

After completion of study treatment, patients are followed up at 1 week, 1 month, and every 3 months for 2 years, every 6 months for 3 years and annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Male age >= 18 years
* Karnofsky performance status > 70%
* Expected survival of at least 3 years
* Informed consent signed by the subject
* PSA blood test within 60 days prior to registration
* Prostate biopsy with Gleason score and TNM staging within one year prior to registration
* No evidence of metastasis on computed tomography (CT) or magnetic resonance imaging (MRI) of the pelvis within 120 days prior to registration
* No evidence of metastasis on bone scan within 120 days prior to registration
* Within 60 days prior to registration, hematologic minimal values: absolute neutrophil count > 1,500/mm^3
* Within 60 days prior to registration, hematologic minimal values: hemoglobin > 8.0 g/dl
* Within 60 days prior to registration, hematologic minimal values: platelet count > 100,000/mm^3
* Men of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months after completion of treatment
* Histologically proven persistent or recurrent adenocarcinoma of the prostate following prior external beam radiation therapy or brachytherapy
* Prior androgen deprivation or chemotherapy is allowed if discontinued at least 30 days prior to enrollment
* Concurrent disease - patients under treatment for concurrent medical conditions will be eligible for protocol treatment if, in the opinion of the physician responsible for hyperthermia treatment that the concurrent medical condition will neither interfere with the process of the treatment or patient assessments nor add significantly to the risks or complications of the treatment

Exclusion Criteria:

* History of urological surgery or procedures predisposing to genitourinary (GU) complications after radiation, i.e., anastomoses, stricture repair, transurethral resection, etc. (will be determined by radiation oncologist)
* Prior thermal ablative therapy for prostate cancer (e.g. high-intensity focused ultrasound [HIFU] or cryoablation)
* Documented distant metastatic disease
* Patient with other co-morbidities that in the opinion of the treating physician would be a contra-indication to protocol participation (e.g. inflammatory bowel disease)
* Mental incompetence or criminal incarceration

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity defined as >= grade 3 per National Cancer Institute Common Toxicity Criteria version 4 occurring within 90 days of treatment and at least possibly attributed to radiation therapy and/or hyperthermia | Up to 90 days
  Will be computed with the corresponding 90% exact binomial confidence intervals.

SECONDARY OUTCOMES:
Incidence of long-term toxicity associated with combined salvage high dose rate (HDR) brachytherapy and interstitial hyperthermia | Up to 5 years
  Will be computed with the corresponding 90% exact binomial confidence intervals.
Efficacy of combined salvage HDR brachytherapy and interstitial hyperthermia as defined by nadir PSA =< 0.5 mg/ml and freedom from biochemical failure per the Phoenix definition (nadir + 2) | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jessie DiNome, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/